CLINICAL TRIAL: NCT00185328
Title: A Multi-Center, Open-Label, Non-Comparative Study Investigating the Efficacy and Tolerability of Angeliq® in Postmenopausal Thai Women With Vasomotor Symptoms Over Three 28-Day Treatment Cycles
Brief Title: Efficacy and Tolerability of Angeliq in Thai Women
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Medical Affairs Therapeutic Area Head, Bayer Schering Pharma AG
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 91436; 309367
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2008-12-12 (Estimated); Status verified 2008-12

CONDITIONS: Postmenopause
Keywords: Postmenopause
MeSH Terms: interventions — estradiol-drospirenone combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: Estradiol/DRSP (Angeliq, BAY86-4891)

INTERVENTIONS:
Drug: Estradiol/DRSP (Angeliq, BAY86-4891) — 1 tablet of 2 mg drospirenone and 1 mg estradiol, orally administered once daily, over three 28-day treatment cycles

SUMMARY:
To evaluate the safety, tolerability, and efficacy of Angeliq in Thai post menopausal women with hot flushes and other climacteric symptoms.

DETAILED DESCRIPTION:
The study has previously been posted by Schering AG, Germany. Schering AG, Germany has been renamed to Bayer Schering Pharma AG, Germany.

Bayer Schering Pharma AG, Germany is the sponsor of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women with hot flushes

Exclusion Criteria:

* Women with a contraindication for Hormone Replacement Therapy (HRT)

Min Age: 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2005-09; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
The relative change in the frequency of hot flushes | At baseline, week 4, 8, 12

SECONDARY OUTCOMES:
The change in intensity of hot flushes | At baseline, week 4, 8, 12
The relative change in frequency of hot flushes | At baseline, week 4, 8
The change in intensity of hot flushes | At baseline, week 4, 8
The proportions of subjects with urogenital symptoms | At baseline, week 4, 8, 12
Bleeding pattern | At baseline, week 4, 8, 12
Adverse events collection | Collection of AE throughout the study period

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer